CLINICAL TRIAL: NCT00187616
Title: Questioning Patients About Adverse Medical Events: A Randomized Controlled Trial
Brief Title: Questioning Patients About Adverse Medical Events
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: STEPAE-001
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: adverse events; clinical trial methodology
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This trial studies whether 3 different methods of asking patients about adverse medical events in a clinical trial affects the rate of reported side effects.

DETAILED DESCRIPTION:
214 patients involved in a larger randomized controlled trial of the herb, saw palmetto, for benign prostatic hyperplasia were randomly assigned to 3 different methods of adverse event ascertainment after a 1-month placebo run-in visit. Two methods of ascertainment were open ended questions, and 1 was a checklist. Patients were blinded to group assignment, but investigators were aware (single blind). All patients had taken placebo for one month, but had been told it was a study drug (single blind).

ELIGIBILITY:
Inclusion Criteria:

* Male, age > 49, American Urological Association Symptom Index > 8
* Max urine flow rate > 4 and < 15

Exclusion Criteria:

* prior prostate cancer or surgery
* use of medications that affect urination
* severe concomitant illness

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214
Dates: Start 2002-04; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Bent, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States